CLINICAL TRIAL: NCT05906277
Title: Melanoma 4p: Biobanking and New Biomolecular Metrics
Brief Title: Biobanking and New Biomolecular Metrics
Acronym: Melamoma4p
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Istituti Fisioterapici Ospitalieri (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: RS1174/19
Record Dates: First submitted 2023-03-24; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-03

CONDITIONS: Melanoma (Skin); Liquid Biopsy
MeSH Terms: conditions — Melanoma | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: The recruiting of two simultaneous cohorts is scheduled. a) patients of illness onset (Cohort 1); b) patients with locoregional disease and/or metastatic designed for systemic therapies (cohort 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biopsy — Liquid biopsy, re-biopsy, tissue biopsy

SUMMARY:
The goal of this Interventional study aims to apply, in our Institutes, a 4p oncological model i.e. predictive, personalized, of precision and participated (Regina Elena and San Gallicano).

DETAILED DESCRIPTION:
Patients will be recruited with an innovative and systematic scheme: collection and biobanking of biological materials (tissue biopsy, re-biopsy and liquid biopsy) followed by a molecular monitoring thanks to genomic and epigenomic methods. It's an open-ended study. In particular we will try to identify new "actionable" signatures and we will try to insert the patients to innovative clinical trials, thanks to the evaluation of all cases with a Molecular Tumor Board.

The main objectives are:

* Introduce a new methodology to improve and integrate the already existent institutional PDTA
* Evaluate and measure the applicative value
* Establish a biostatistical platform

ELIGIBILITY:
Inclusion Criteria:

* Melanoma affected patients

Exclusion Criteria:

* No patiens affected by other pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Oncology target therapy | 12 months
  Integration between molecular diagnostic and melanoma histopathology: correlation between mutational miRNA/ncRNA profiles and pathological staging parameters.
Oncology target therapy | 12 months
  Correlation between molecular diagnostic and imaging non-invasive instrumental diagnostic
Oncology target therapy | 12 months
  Correlation between molecular diagnostic and dermatologic clinical diagnostic; integration of liquid biopsy during oncologic ambulatorial follow-up; lead time of relapse.
Oncology target therapy | 12 months
  Complement to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- IRE, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided